CLINICAL TRIAL: NCT03083730
Title: Impact of Narrowband UVB Phototherapy on Systemic Inflammation in Patients With Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Principal Investigator, James G. Krueger, MD, PhD, Professor, Rockefeller University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PBR-0933
Record Dates: First submitted 2017-03-01; First posted 2017-03-20 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Eczema; Systemic Inflammation; UVB Phototherapy
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atopic Dermatitis Cohort (Experimental): Narrow band UVB treatment (NB-UVB) NB-UVB light treatment 3x/week for 12 weeks (36 visits)
  Healthy Control Cohort will be obtained to take baseline blood work as a reference value for baseline expression of blood markers.
  Interventions: Other: Narrow band UVB treatment (NB-UVB)

INTERVENTIONS:
Other: Narrow band UVB treatment (NB-UVB) — NB-UVB light treatment NB-UVB light treatment for 3x/week for 12 weeks (36 visits)

SUMMARY:
Atopic dermatitis (eczema) is a chronic inflammatory disease that causes significant morbidity and is now known to be associated with cardiovascular disease. Research such as this will add to the understanding of the skin as a contributor to systemic inflammation, and it is important to clarify whether skin-only treatment can alleviate systemic inflammation, and potentially influence cardiovascular risk factors.

DETAILED DESCRIPTION:
Globally, the leading cause of death is cardiovascular disease, which is often linked to chronic inflammation.

Recently, it has been shown that atopic dermatitis (AD), the most common chronic inflammatory skin disease, shows increases in inflammatory and cardiovascular risk markers in patient blood (proteins, microparticles, circulating inflammatory cells). Consistently, it has been demonstrated that atopic dermatitis is associated with increased cardiovascular disease. Whether these increases in inflammatory and/or cardiovascular risk markers in the peripheral blood are due to skin inflammation, or due to other body sources (e.g. lung, lymphatic system) is unknown.

To investigate whether some (or all) risk proteins present in patient blood are produced in inflamed skin, the investigators want to treat patients suffering from moderate-to-severe AD with ultra-violet light B (UVB) therapy, as this therapy is thought to be an exclusive skin treatment, without direct systemic effects. This notion is corroborated by the fact that only skin regions directly treated with UVB light, and not covered skin regions, respond to phototherapy.

Ultra-violet light B (UVB) therapy has been used by dermatologists to treat AD for decades, and in the 1990ies, narrow band-UVB (NB-UVB) wavelengths (311-312nm) were found to have the best treatment effects. This is a safe and effective therapy for the majority of patients, with the main drawback being that it is inconvenient, as patients need to attend the clinic three times a week for at least 8 weeks. The mechanism of action appears to include killing of skin immune cells, and it also appears to down regulate inflammatory molecules such as IFNg, IL-12 and IL-23. However, a systematic study of the impact of NBUVB on blood biomarkers has never been performed. In this study, participants will be treated with an appropriate dose of NB-UVB three times a week for up to 12 weeks or a total of 36 treatments, and blood will be drawn to assess inflammatory and cardiovascular risk markers (proteins, microparticles, circulating blood cells). Results will be compared to levels in blood from healthy control participants. This study could lead to a new understanding on the role of the skin as a source of systemic inflammation, which would help to guide future treatment approaches for this debilitating, chronic skin disease.

ELIGIBILITY:
Inclusion Criteria:

ATOPIC DERMATITIS COHORT

1. At least 18 years of age
2. >10% body surface affected
3. History of atopic dermatitis for at least 3 years (as per patient history)

HEALTHY CONTROL COHORT

1. At least 18 years of age

Exclusion Criteria:

ATOPIC DERMATITIS COHORT

1. Unstable or persistent asthma (mild, moderate, or severe), i.e. all forms of allergic asthma that are other than intermittent asthma. Intermittent asthma is allowed: Difficulty breathing, wheezing, chest tightness, and coughing occur on fewer than 2 days a week, do not interfere with normal activities, and nighttime symptoms occur on fewer than 2 days a month.
2. Use of topical glucocorticosteroids or other immunosuppressive topical therapy within 1 week of treatment initiation. Emollients are allowed.
3. Untreated skin malignancy
4. Use of systemic anti-inflammatory medication in the last 4 weeks for more than 3 days
5. Known photosensitivity: Hypersensitivity to sunlight or UVB light of any type or photosensitizing medication
6. History of Lupus, Polymorphic light eruption (PMLE), or any disease known to be worsened by UV light exposure
7. History of melanoma
8. History, physical, social or lab findings suggestive of any medical or psychological condition that would, in the opinion of the PI make the candidate ineligible for the study

HEALTHY CONTROL COHORT

1. self-reported chronic inflammatory diseases (IBD, rheumatoid arthritis, collagenoses, chronic inflammatory skin disease, Atopic Dermatitis, autoimmune or autoinflammatory disease, active tuberculosis, chronic infectious disease such as HIV and hepatitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Systemic Inflammation | 12 weeks
  Change from baseline of inflammatory and cardiovascular risk proteins in serum of atopic dermatitis patients during treatment with NB-UVB.

SECONDARY OUTCOMES:
Microparticles | 12 weeks
  Change from baseline of microparticles in the peripheral blood of Atopic Dermatitis patients treated with NB-UVB
PBMC activation markers | 12 weeks
  Change from baseline in PBMC activation markers in the peripheral blood of Atopic Dermatitis patients treated with NBUVB
Disease Scores (SCORAD) | 12 weeks
  Change from baseline in clinical skin disease scores (SCORAD) in Atopic Dermatitis patients treated with NBUVB
Disease Scores (EASI) | 12 weeks
  Change from baseline in clinical skin disease scores (EASI) in Atopic Dermatitis patients treated with NBUVB
Disease Scores (IGA) | 12 weeks
  Change from baseline in clinical skin disease scores (IGA) in Atopic Dermatitis patients treated with NBUVB
Comparison to healthy controls | 12 weeks
  Number of markers significantly increased/decreased compared to healthy control samples, and their change during treatment
Correlation with skin markers | 12 weeks
  Correlation of inflammatory markers between serum and skin before and after NB-UVB treatment

CONTACTS AND LOCATIONS:
Overall Officials: Patrick M Brunner, MD, Principal Investigator — The Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Silverberg JI, Greenland P. Eczema and cardiovascular risk factors in 2 US adult population studies. J Allergy Clin Immunol. 2015 Mar;135(3):721-8.e6. doi: 10.1016/j.jaci.2014.11.023. Epub 2015 Jan 8. PMID 25579484
- [Background] Hjuler KF, Bottcher M, Vestergaard C, Deleuran M, Raaby L, Botker HE, Iversen L, Kragballe K. Increased Prevalence of Coronary Artery Disease in Severe Psoriasis and Severe Atopic Dermatitis. Am J Med. 2015 Dec;128(12):1325-34.e2. doi: 10.1016/j.amjmed.2015.05.041. Epub 2015 Jun 18. PMID 26093174
- [Background] Erbel C, Chen L, Bea F, Wangler S, Celik S, Lasitschka F, Wang Y, Bockler D, Katus HA, Dengler TJ. Inhibition of IL-17A attenuates atherosclerotic lesion development in apoE-deficient mice. J Immunol. 2009 Dec 15;183(12):8167-75. doi: 10.4049/jimmunol.0901126. PMID 20007582
- [Background] Czarnowicki T, Malajian D, Shemer A, Fuentes-Duculan J, Gonzalez J, Suarez-Farinas M, Krueger JG, Guttman-Yassky E. Skin-homing and systemic T-cell subsets show higher activation in atopic dermatitis versus psoriasis. J Allergy Clin Immunol. 2015 Jul;136(1):208-11. doi: 10.1016/j.jaci.2015.03.032. Epub 2015 May 1. No abstract available. PMID 25936564
- [Background] Tamagawa-Mineoka R, Katoh N, Ueda E, Masuda K, Kishimoto S. Platelet-derived microparticles and soluble P-selectin as platelet activation markers in patients with atopic dermatitis. Clin Immunol. 2009 Jun;131(3):495-500. doi: 10.1016/j.clim.2009.01.006. Epub 2009 Feb 13. PMID 19217350
- [Background] Ungar B, Garcet S, Gonzalez J, Dhingra N, Correa da Rosa J, Shemer A, Krueger JG, Suarez-Farinas M, Guttman-Yassky E. An Integrated Model of Atopic Dermatitis Biomarkers Highlights the Systemic Nature of the Disease. J Invest Dermatol. 2017 Mar;137(3):603-613. doi: 10.1016/j.jid.2016.09.037. Epub 2016 Nov 4. PMID 27825969